CLINICAL TRIAL: NCT03325283
Title: Cerebral Protection in Transcatheter Aortic Valve Replacement
Brief Title: The PROTEMBO SF Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Protembis GmbH (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CIP_00104, Rev 02, 23 May 2017
Record Dates: First submitted 2017-10-13; First posted 2017-10-30 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Aortic Stenosis
Keywords: stroke prevention; embolic protection; cognition
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: Human patients indicated for transcatheter aortic valve replacement
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Protembo device treatment (Experimental): Patients who consent to participate in the PROTEMBO SF Trial and in whom the ProtEmbo Cerebral Protection System is used or is attempted to be used.
  Interventions: Device: ProtEmbo Cerebral Protection System

INTERVENTIONS:
Device: ProtEmbo Cerebral Protection System — A catheter-based embolic deflection device will be positioned in the arch of the aorta to prevent debris liberated during the TAVR procedure from entering the three major vessels of the aortic arch.

SUMMARY:
The PROTEMBO SF Trial is a prospective, observational, multi-center, intention-to-treat study of the safety and feasibility of the ProtEmbo Cerebral Protection System in subjects with severe symptomatic native aortic valve stenosis indicated for TAVR.

DETAILED DESCRIPTION:
The PROTEMBO SF Trial is a prospective, single arm, observational, multi-center, intention-to-treat study of the safety and feasibility of the ProtEmbo Cerebral Protection System in subjects with severe symptomatic native aortic valve stenosis indicated for TAVR.

ELIGIBILITY:
Inclusion Criteria:

1. Approved indications for commercially available transcatheter aortic valves by transfemoral route. Refer to the selected valve IFU for additional details.
2. Compatible left subclavian artery (≥ 4 mm diameter) without significant stenosis (> 70%) and distance between the origin of left subclavian artery and valve plain is ≥ 90mm as determined by Multi-Slice Computed Tomography (MSCT) scan or equivalent imaging modality.
3. The subject and the treating physician agree that the subject will undergo the scheduled pre-procedural testing and return for all required post-procedure follow-up visits.
4. The subject has been informed of the nature of the trial, agrees to its provisions and has provided written informed consent as approved by the national or local regulatory authorities of the respective clinical site.
5. Subject is a minimum of 18 years of age.

Exclusion Criteria:

1. Left upper limb vasculature precluding 6Fr sheath (radial or brachial access).
2. Inadequate circulation to the left extremity as evidenced by signs of artery occlusion (modified Allen's test) or absence of radial/ brachial pulse.
3. Hemodialysis shunt, graft, or arterio-venous fistula involving the upper extremity vasculature.
4. TAVR conducted via other than transfemoral access (subclavian, axillar, transapical, transaortic, carotid or transcaval).
5. Evidence of an acute myocardial infarction ≤ 1 month before the intended treatment.
6. Aortic valve is a congenital unicuspid or bicuspid valve.
7. Mixed aortic valve disease (aortic stenosis and aortic regurgitation with predominant aortic regurgitation >3+).
8. Any therapeutic invasive cardiac procedure resulting in a permanent implant that is performed within 30 days of the index procedure (unless part of planned strategy for treatment of concomitant coronary artery disease).
9. Pre-existing prosthetic heart valve in any position, prosthetic ring, or severe (greater than 3+) mitral insufficiency.
10. Blood dyscrasias as defined: Leukopenia, acute anemia, thrombocytopenia, history of bleeding diathesis or coagulopathy.
11. Hemodynamic instability requiring inotropic support or mechanical heart assistance.
12. Need for emergency surgery for any reason.
13. Severe hypertrophic cardiomyopathy with or without obstruction.
14. Severe ventricular dysfunction with LVEF ≤30%.
15. Echocardiographic evidence of intracardiac or aortic mass, thrombus, or vegetation.
16. Symptomatic or asymptomatic severe (≥ 70%) occlusive carotid disease requiring concomitant CEA/ stenting.
17. Subject has undergone carotid stenting or carotid endarterectomy within the previous 6 weeks.
18. Active peptic ulcer or upper GI bleeding within the prior 3 months.
19. A known hypersensitivity or contraindication to aspirin, heparin, ticlopidine, or clopidogrel, device component material, or sensitivity to contrast media, which cannot be adequately pre-medicated.
20. Recent (within 6 months) CVA or a TIA.
21. Renal insufficiency (creatinine > 3.0 mg/ dL or GFR < 30) and/ or renal replacement therapy at the time of screening.
22. Life expectancy < 12 months due to non-cardiac comorbid conditions.
23. Subjects in whom anti-platelet and/ or anticoagulant therapy is contraindicated, or who will refuse transfusion.
24. Subjects who have active bacterial endocarditis or other active infections.
25. Currently participating in an investigational drug or another device study.
26. Subjects who have a planned treatment with any other investigational device or procedure during the study follow-up period (30 days).
27. Subjects with planned concomitant surgical or transcatheter ablation for Atrial fibrillation during the study follow-up period (30 days).
28. Any subject with a balloon valvuloplasty (BAV) within 30 days of the procedure.
29. Subject is a woman of child bearing age.
30. Patient with Heparin-Induced Thrombocytopenia Syndrome.
31. Inner diameter of aortic arch is less than 25mm.
32. Type I Aortic Arch: Distance of the origin of the innominate artery from the top of aortic arch is less than one times the diameter of left common carotid artery.
33. Brachiocephalic trunk originating from the aortic arch that splits into the bilateral subclavian arteries and a bicarotid trunk (Origin D).

Neurological:

1. Subject has active major psychiatric disease.
2. Subject has severe visual, auditory, or learning impairment and is unable to comprehend English or local language and therefore unable to be consented for the study.
3. Subjects with neurodegenerative or other progressive neurological disease or history of significant head trauma followed by persistent neurologic defaults or known structural brain abnormalities.

Angiographic:

1. Excessive tortuosity in the left radial/ brachial/subclavian artery preventing ProtEmbo System access and insertion.
2. Subject whose left radial/ brachial/ subclavian artery reveals significant stenosis, calcification, ectasia, dissection, or aneurysm.

Magnetic Resonance Imaging:

1. Subject Body Mass Index (BMI) precluding imaging in scanner.
2. Contraindications to MRI (subjects with any implantable temporary or permanent pacemaker or defibrillator, metal implants in field of view, metallic fragments, clips, or devices in the brain or eye before TAVR procedure).
3. Patients who have a high risk of complete AV block after TAVR, with the need of permanent pacemaker (e.g. patients with pre-existing bifascicular block or complete right bundle branch block plus any degree of AV block).
4. Planned implantation of a pacemaker or defibrillator implantation within the first 7 days after TAVR.
5. Claustrophobia precluding MRI scanning.
6. No scanner hardware, software, coil or protocol changes should occur during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-08-09 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Procedural success | 1 day
  defined as successful access, delivery to, deployment within, and retrieval of the ProtEmbo System from the aortic arch as well as adequate coverage of side branch vessels and maintenance of position for duration of the TAVR procedure.
In-hospital procedural safety up to 7 days | 7 days
  defined as occurrence of all Major Adverse Cardiac and Cerebrovascular Events (MACCEs) defined by the Valve Academic Research Consortium (VARC-2) criteria, including device-related safety outcomes (peri-procedural rates of TIA, all-cause mortality, all stroke (disabling and non-disabling), life-threatening (or disabling) bleeding, acute kidney injury (stage 2 or 3), major vascular complications and other device related complications).
Stroke severity | 3 days
  quantified according to the National Institutes of Health Stroke Scale (NIHSS) score at day 3 (±2).
Stroke severity | 30 days
  quantified according to the National Institutes of Health Stroke Scale (NIHSS) score at 30 days (±7).
Occurrence of Serious Adverse Events | 3 days
  as defined by ISO 14155 up to 3 (±2) days or discharge (whichever is later) and 30 days (±7).
Occurrence of Serious Adverse Events | 30 days
  as defined by ISO 14155 at 30 days (±7).

SECONDARY OUTCOMES:
Frequency of new cerebral lesions | 3 days
  defined by diffusion weighted magnetic resonance imaging (DW-MRI) prior to discharge at day 3 (±2) compared to baseline and/ or historical control group;
Number of new cerebral lesions | 3 days
  defined by diffusion weighted magnetic resonance imaging (DW-MRI) prior to discharge at day 3 (±2) compared to baseline and/ or historical control group;
Volume of new cerebral lesions | 3 days
  defined by diffusion weighted magnetic resonance imaging (DW-MRI) prior to discharge at day 3 (±2) compared to baseline and/ or historical control group;
Frequency of new cerebral lesions | 30 days
  defined by Diffusion weighted- and FLAIR-MRI sequence at 30 days (±7 days).
Number of new cerebral lesions | 30 days
  defined by Diffusion weighted- and FLAIR-MRI sequence at 30 days (±7 days).
Volume of new cerebral lesions | 30 days
  defined by Diffusion weighted- and FLAIR-MRI sequence at 30 days (±7 days).
Cognitive function | 30 days
  defined as change in neurocognitive testing at 30 (+/- 7) days post-procedure using MoCA post-procedure compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: James C. Leiter, M.D., Study Director — Avania
Locations (2):
- Department of Cardiology Galway University Hospital and SAOLTA Healthcare Group, Galway, County Galway, Ireland
- Pauls Stradins Clinical University Hospital, Riga, Latvia

IPD SHARING:
Plan to Share IPD: No